CLINICAL TRIAL: NCT00476710
Title: Effects of Colesevelam HCl On Bile Acid Pools And Kinetic Parameters in Normal Subjects, Subjects With Impaired Glucose Tolerance, And Subjects With Type 2 Diabetes Mellitus
Brief Title: Effects of Colesevelam HCl On Bile Acid Kinetics
Status: Completed | Type: Observational
Sponsor: KineMed (Industry)
Collaborators: Daiichi Sankyo (Industry); University Medical Center Groningen (Other); Diabetes & Glandular Disease Research Associates (Unknown)
Responsible Party: Sponsor
Other Study IDs: KM-11B
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus; Impaired Glucose Tolerance
Keywords: Type 2 diabetes mellitus; Bile acid; Stable isotope; Colesevelam HCl; Impaired Glucose Tolerance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal Glucose Metabolism: Overweight and obese individuals that have normal glucose metabolism and their response to Colesevelam HCl
  Interventions: Drug: Colesevelam HCl
- Impaired Glucose Tolerance: Overweight and obese individuals that have impaired glucose tolerance and their response to Colesevelam HCl
  Interventions: Drug: Colesevelam HCl
- Frank type 2 diabetes: Overweight and obese individuals that have frank type 2 diabetes and their response to Colesevelam HCl
  Interventions: Drug: Colesevelam HCl

INTERVENTIONS:
Drug: Colesevelam HCl

SUMMARY:
This project will compare the amount of bile acids and their kinetics in overweight and obese people with normal glucose metabolism, impaired glucose tolerance and frank type 2 diabetes. We hypothesize that bile acids will behave differently in these groups. We will also explore the effects of Colesevelam HCl, a medicine that lowers LDL cholesterol by binding bile acids, on bile acids in those groups. We hypothesize the drug may have different actions on bile acids in subjects with different degrees of abnormal glucose metabolism.

DETAILED DESCRIPTION:
Bile acids, which are synthesized from cholesterol in the liver, play a key role in digestion as they solubilize dietary lipids and aid their absorption in the digestive tract. While for many years bile acids have been characterized by this digestive role, recent research indicates that bile acids play other important roles. Because bile acids have been shown to act in signaling pathways that affect metabolism, there has been renewed interest in investigations of their effects. This study explores potential differences in bile acid kinetics based on insulin resistance or type 2 diabetes at baseline.

Colesevelam HCl is a bile acid sequestrant, which in addition to its primary role in lowering serum LDL-C levels, has secondarily been implicated in lowering blood glucose levels. This study explores the relationship between insulin resistance and type 2 diabetes and changes in bile acid pool sizes and kinetics with colesevelam treatment. Isotopically labeled bile acids will be administered to subjects before and after treatment with colesevelam and comparisons will be made in bile acid pool size, fractional turnover rate, and synthesis rate in the three study groups.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* BMI 25-35 kg/m^2, inclusive
* Normal liver and thyroid function
* No history of liver, biliary, or intestinal disease

Diabetic Subjects

* Diagnosed Type 2 Diabetes Mellitus
* HbA1C = 6.7-10%

Normal Subjects

* 2 hr OGTT glucose < 140 mg/dL
* fasting glucose < 100 mg/dL
* TG < 150 mg/dL
* HDL cholesterol >= 40 mg/dL

Impaired Glucose Tolerance Subjects

* 2 hr OGTT glucose >= 140 and < 200 mg/dL

Exclusion Criteria:

* T1DM or history of diabetic ketoacidosis
* treatment with blood pressure lowering therapy that has not been stable for three months before screening
* colesevelam HCl, cholestyramine, or colestipol treatment for hyperlipidemia within the last three months
* treatment with thiazolidinedione (TZD) at any time
* treatment with insulin within past 6 months
* treatment with antibiotics within last 3 months
* extreme sportsmen
* treatment with medication affecting liver or intestinal function within the last 3 months
* allergic or toxic rxn to colesevelam HCl
* history of dysphagia, swallowing disorders, or intestinal motility disorder
* Serum Triglycerides > 500 mg/dL at visit 1
* Serum LDL-C < 60 mg/dL at visit 1
* any condition or therapy investigator believes not in subjects best interest
* use of any investigational drug within 30 days before screening
* chronic treatment with oral corticosteroids at any time or acute treatment within last three months
* hyperthyroidism or treatment with thyroid hormone/levothyroxine

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: overweight and obese people with normal glucose metabolism, impaired glucose tolerance and frank type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2007-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Bile Acid Pool Size and Kinetic Parameters | 60 days of treatment

SECONDARY OUTCOMES:
Resting Metabolic Rate | 60 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Murphy, MD, Principal Investigator — KineMed, Inc.; Folkert Kuipers, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- Diabetes & Glandular Disease Research Associates, Inc., San Antonio, Texas, United States

REFERENCES:
- [Background] Grundy SM, Ahrens EH Jr, Salen G. Interruption of the enterohepatic circulation of bile acids in man: comparative effects of cholestyramine and ileal exclusion on cholesterol metabolism. J Lab Clin Med. 1971 Jul;78(1):94-121. No abstract available. PMID 5569253
- [Background] Shepherd J, Packard CJ, Bicker S, Lawrie TD, Morgan HG. Cholestyramine promotes receptor-mediated low-density-lipoprotein catabolism. N Engl J Med. 1980 May 29;302(22):1219-22. doi: 10.1056/NEJM198005293022202. PMID 7366673
- [Background] Zieve FJ, Kalin MF, Schwartz SL, Jones MR, Bailey WL. Results of the glucose-lowering effect of WelChol study (GLOWS): a randomized, double-blind, placebo-controlled pilot study evaluating the effect of colesevelam hydrochloride on glycemic control in subjects with type 2 diabetes. Clin Ther. 2007 Jan;29(1):74-83. doi: 10.1016/j.clinthera.2007.01.003. PMID 17379048
- [Background] Abrams JJ, Ginsberg H, Grundy SM. Metabolism of cholesterol and plasma triglycerides in nonketotic diabetes mellitus. Diabetes. 1982 Oct;31(10):903-10. doi: 10.2337/diab.31.10.903. PMID 6759223
- [Background] Andersen E, Karlaganis G, Sjovall J. Altered bile acid profiles in duodenal bile and urine in diabetic subjects. Eur J Clin Invest. 1988 Apr;18(2):166-72. doi: 10.1111/j.1365-2362.1988.tb02408.x. PMID 3133222
- [Background] Bennion LJ, Grundy SM. Effects of diabetes mellitus on cholesterol metabolism in man. N Engl J Med. 1977 Jun 16;296(24):1365-71. doi: 10.1056/NEJM197706162962401. PMID 870827
- [Background] Hulzebos CV, Renfurm L, Bandsma RH, Verkade HJ, Boer T, Boverhof R, Tanaka H, Mierau I, Sauer PJ, Kuipers F, Stellaard F. Measurement of parameters of cholic acid kinetics in plasma using a microscale stable isotope dilution technique: application to rodents and humans. J Lipid Res. 2001 Nov;42(11):1923-9. PMID 11714862
- [Derived] Brufau G, Stellaard F, Prado K, Bloks VW, Jonkers E, Boverhof R, Kuipers F, Murphy EJ. Improved glycemic control with colesevelam treatment in patients with type 2 diabetes is not directly associated with changes in bile acid metabolism. Hepatology. 2010 Oct;52(4):1455-64. doi: 10.1002/hep.23831. PMID 20725912
- See also: Related Info — http://www.kinemed.com